CLINICAL TRIAL: NCT03308474
Title: Clinical Research Platform for Molecular Testing, Treatment and Outcome of Patients With Multiple Myeloma (Myeloma Registry Platform; MYRIAM)
Brief Title: Myeloma Registry Platform (MYRIAM)
Acronym: MYRIAM
Status: Recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Deutsche Studiengruppe Multiples Myelom (DSMM) (Unknown)
Responsible Party: Sponsor
Other Study IDs: iOM-060331
Record Dates: First submitted 2017-09-25; First posted 2017-10-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Routine care as per site standard. — Physician's choice according to patient's needs.

SUMMARY:
The purpose of the project is to set up a national, prospective, longitudinal, multicenter cohort study with associated satellites, a tumor registry platform, to document uniform data on characteristics, molecular diagnostics, treatment and course of disease, to collect patient-reported outcomes and to establish a decentralized biobank for patients with Multiple Myeloma in Germany.

DETAILED DESCRIPTION:
MYRIAM is a national, observational, prospective, longitudinal, multicenter cohort study (tumor registry platform) with the purpose to record information on the antineoplastic treatment of multiple myeloma in Germany. The registry will follow patients for up to five years. It will identify common therapeutic sequences and changes in the treatment of the disease. At inclusion, data in patient characteristics, comorbidities, tumor characteristics and previous treatments are collected. During the course of observation data on all systemic treatments, radiotherapies, surgeries, and outcome are documented.

Health-realted quality of life in patients with multiple myeloma (MyLife) will be evaluated for up to five years.

ELIGIBILITY:
Inclusion Criteria:

* MM requiring systemic (first-, second- or third-line) treatment (closed for first-line / second-line recruitment)
* Age ≥ 18 years
* Written informed consent

  * Patients participating in the PRO satellite: signing of informed consent and completion of baseline questionnaire before, but not more than eight weeks before the start of respective systemic treatment
  * Patients not participating in the PRO satellite: signing of informed consent not later than four weeks after start of respective treatment, and not more than eight weeks before the start of respective systemic treatment
* Sufficient German language skills for participation in the PRO satellite

Exclusion Criteria:

* No systemic therapy for myeloma
* Patients already enrolled in studies that prohibit any participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with multiple myeloma (MM) requiring systemic treatment
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2017-09-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Course of treatment (treatment reality) | 5 years per patient
  Documentation of anamnestic data and therapy sequences

SECONDARY OUTCOMES:
Best Response | 5 years per patient
  Documentation of response rates per line of treatment.
Progression-free survival | 5 years per patient
  Documentation of progression-free survival per line of treatment.
Overall survival | 5 years per patient
  Documentation of overall survival time.
Health-related quality of life (Patient-reported outcome) | 5 years per patient
  EORTC QLQ-C30 core questionnaire.
Myeloma-specific health-related quality of life (Patient-reported outcome) | 5 years per patient
  EORTC QLQ-MY20, the myeloma specific module.
Quality of life (Patient-reported outcome) | 5 years per patient
  Brief Pain Inventory (BPI)

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Einsele, Prof MD, Study Chair — Wuerzburg University Hospital; Monika Engelhardt, Prof MD, Study Chair — Universitätsklinikum Freiburg; Tobias Dechow, Prof MD, Study Chair — Onkologie Ravensburg; Wolfgang Knauf, Prof MD, Study Chair — Centrum für Hämatologie und Onkologie Bethanien; Norbert Marschner, MD, Study Chair — Praxis für interdisziplinäre Onkologie & Hämatologie
Locations (1):
- Multiple sites all over germany, Multiple Sites, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Engelhardt M, Ihorst G, Singh M, Rieth A, Saba G, Pellan M, Lebioda A. Real-World Evaluation of Health-Related Quality of Life in Patients With Multiple Myeloma From Germany. Clin Lymphoma Myeloma Leuk. 2021 Feb;21(2):e160-e175. doi: 10.1016/j.clml.2020.10.002. Epub 2020 Oct 24. PMID 33218965